CLINICAL TRIAL: NCT00098618
Title: A Phase 2 Study Of BAY 43-9006 In Combination With Interferon Alfa-2b In Metastatic Renal Cell Cancer
Brief Title: Sorafenib and Interferon Alfa in Treating Patients With Locally Advanced or Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02638; 6258-04-9R0; NCI-6553; CDR0000398171; U01CA099118 (NIH)
Record Dates: First submitted 2004-12-07; First posted 2004-12-08 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Clear Cell Renal Cell Carcinoma; Papillary Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib; Interferon-alpha; Interferon Alfa-n3; Introns; Interferon alpha-2

ARMS (1):
- Treatment (sorafenib tosylate and recombinant interferon alfa) (Experimental): Patients receive oral sorafenib twice daily and interferon alfa subcutaneously three times a week for 8 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: sorafenib tosylate; Biological: recombinant interferon alfa; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Biological: recombinant interferon alfa — Given orally
  Other Names: Alferon N; alpha interferon; IFN-A; Intron A; Roferon-A
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for their growth or by blocking blood flow to the tumor. Interferon alfa may interfere with the growth of tumor cells and slow the growth of kidney cancer. Sorafenib may help interferon alfa kill more tumor cells by making tumor cells more sensitive to the drug. Giving sorafenib together with interferon alfa may kill more tumor cells. This phase II trial is studying how well giving sorafenib with interferon alfa works in treating patients with locally advanced or metastatic kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility and tolerability of sorafenib and interferon alfa in patients with locally advanced or metastatic renal cell carcinoma.

II. Determine the response rate (complete response and partial response) in patients treated with this regimen.

SECONDARY OBJECTIVES:

I. Determine the progression-free survival and response duration of patients treated with this regimen.

II. Correlate changes in laboratory parameters with response in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily and interferon alfa subcutaneously three times a week for 8 weeks. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

Patients with stable or responding disease are followed every 3 months for 2 years, every 6 months for 2 years, and then annually for 1 year or until disease progression.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 10 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed renal cell carcinoma

  * Locally advanced or metastatic disease
  * All histologic subtypes allowed
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm by spiral CT scan
* No known brain metastases or leptomeningeal disease
* Performance status - ECOG 0-2
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No bleeding diathesis
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 60 mL/min
* No uncontrolled hypertension
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No history of sensitivity to E. coli-derived products
* No history of severe depression
* No active infection requiring antibiotics
* No seizure disorder requiring antiepileptic medication
* No medical condition likely to require systemic corticosteroids
* No autoimmune disorder that could result in life-threatening complications
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No more than 1 prior biologic response modifier regimen
* At least 4 weeks since prior biologic response modifiers
* No prior interferon alfa
* No prior chemotherapy
* At least 4 weeks since prior radiotherapy to non-index lesions

  * Prior radiotherapy to index lesion allowed provided irradiated lesion progressed ≥ 20% in diameter
* At least 2 weeks since prior major surgery
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapeutic anticoagulation therapy

  * Concurrent prophylactic anticoagulation, such as low-dose warfarin, for venous or arterial access device allowed provided PT, PTT, and INR are normal
* No other concurrent investigational agents
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-10; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Overall response rate (CR+PR) using RECIST criteria | Up to 5 years
  CR+PR rate will be calculated with exact 90% confidence intervals.
Grade 3+ toxicities assessed using NCI CTCAE version 3.0 | Up to 5 years
  Toxicities will be tabulated by type and grade. Toxicity rates will be calculated with exact 90% confidence intervals.
Progression-free survival | Up to 5 years
  Kaplan-Meier curves will be used.
Overall survival | Up to 5 years
  Kaplan-Meier curves will be used.
Duration of response | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented , assessed up to 5 years
  Kaplan-Meier curves will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel George, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States